CLINICAL TRIAL: NCT03721458
Title: Whole Genome Sequencing in the Neonatal Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, James Broach, Director of the Institute for Personalized Medicine, Milton S. Hershey Medical Center
Other Study IDs: 00007970
Record Dates: First submitted 2018-04-04; First posted 2018-10-26 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Genetic Diseases, Inborn
MeSH Terms: conditions — Genetic Diseases, Inborn | interventions — Base Sequence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Sequence — Potentially identifying genetic defects that could have clinical significance

SUMMARY:
This research is being done to see if whole genome sequencing (WGS) improves the diagnosis of patients in the NICU. Using WGS in this way, which is relatively new, researchers at Penn State College of Medicine will look at approximately 5000 genes that are known to be associated with genetic diseases to see if the neonatal patient has a known disease causing mutation. Comparing the parents' DNA with the child's will help the investigators better understand the child's DNA.

DETAILED DESCRIPTION:
1.0 Objectives

1.1 Study Objectives The goal of this research project is to assess the potential for applying whole genome sequencing (WGS) as a diagnostic tool in the neonatal intensive care unit. Newborn children who require treatment in the neonatal intensive care unit (NICU) often suffer from genetic defects, the nature of which is difficult to diagnose. The investigators currently know of more than 5000 genes in which mutations may cause diseases that can affect newborn children, so determining which one is responsible for a new neonatal patient's disease is daunting. However, many of these diseases can be effectively treated if they are diagnosed in a timely fashion. The investigators propose to use new sequencing instrumentation coupled with rapid analytical tools to sequence NICU patients along with both parents to identify whether a patient carries a de novo mutation or compound heterozygous variants in one of the known disease genes. If so, the mutation will be confirmed in an in-house CLIA laboratory and the results provided within 72 hours to attending neonatologists to inform treatment decisions.

1.2 Primary Study Endpoints

The primary goal of this protocol will be an assessment of the degree to which WGS improves diagnosis of patients admitted to the NICU. The investigators propose to perform sequencing on approximately 50 patients over the course of this project. The investigators will evaluate on an ongoing basis the success rate for identifying clinically actionable genetic defects in the selected patients, particularly as that would inform the initial selection criteria used to enroll the patient. This information will be useful to determine whether such sequencing efforts can improve the outcome of NICU patients and which class of patients are most likely to benefit from the procedure.

1.3 Secondary Study Endpoints

A second goal will be an assessment of the effectiveness of targeted sequencing of the whole exome or a panel of 5000 genes in identifying the genetic defects revealed by whole genome sequencing and the relative cost in money and time of the various approaches. This could yield a significantly more efficient and cost effect method over that currently described elsewhere.

Finally, the investigators propose to use the data to begin to develop a cost-benefit analysis of WGS in the NICU. The investigators will assess the extent to which WGS provided a diagnosis distinct from that initially proposed by the neonatologists and the extent to which that change in diagnosis altered the treatment regimen. If the novel diagnosis did, in fact, alter treatment, The investigators would use historical data to assess the degree to which that altered treatment affected the number of days the patient remained in the NICU. The investigators can then estimate the cost savings/loss as the number of NICU days saved times the cost per day of NICU residence versus the cost of performing the sequencing over the entire cohort of sequenced patients. While this is not as rigorous as a randomized clinical trial, it would point to whether this is a methodology worth exploring in more depth.

ELIGIBILITY:
Child:Inclusion Criteria:

1. Age: ≤ 180 days
2. Sex: male or female
3. Admitted to the Hershey Medical Center NICU with a clinical presentation consistent with a genetic disease, e.g. congenital malformations, metabolic disorder, uncontrolled seizures or unexplained abnormal neurological findings.
4. Both Biological Parents are involved in the study

Child:Exclusion Criteria:

1. Age: > 180 days
2. Known genetic mutation.

Biological Parents : Inclusion Criteria

1. Age: ≥18 years
2. Both biological parents must be willing to participate in the research.
3. Fluent in written and spoken English.

Biological Parents: Exclusion Criteria

1. Age: <18 years
2. Prisoner
3. Cognitive impairment

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient is admitted to the NICU, evaluated by the clinical staff, recommended for participation in this study and consented.
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Diagnosis success rate | 1-2 years
  The investigator will determine the percent of patients for which sequencing provided a correct genetic disease diagnosis, relative to that obtained by standard clinical evaluation.

SECONDARY OUTCOMES:
Effectiveness of exome sequencing relative to whole genome sequencing. | 1-2 years
  The investigators will determine whether whole exome sequencing identifies all the genetic disease diagnoses identified by whole genome sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: James Broach, PhD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States